CLINICAL TRIAL: NCT04913285
Title: A Phase 1/1b Open-label, Multicenter Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of KIN-2787 in Participants With BRAF and/or NRAS Mutation-positive Solid Tumors.
Brief Title: A Study to Evaluate KIN-2787 in Participants With BRAF and/or NRAS Mutation Positive Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KN-8701; KIN 2787CI101 (Other: Pierre Fabre Medicament)
Record Dates: First submitted 2021-05-18; First posted 2021-06-04 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor, Adult; Non-small Cell Lung Cancer; Melanoma
Keywords: BRAF inhibitor; BRAF; pan-RAF; pan-RAF inhibitor; RAF1; ARAF; BRAF alteration; BRAF Class II; BRAF Class III; V600; tumor growth inhibitor (TGI); melanoma; NSCLC; solid tumor; targeted therapy; BRAF Class I; NRAS; Metastatic; Unresectable; CRC; ATC; Colon; Thyroid; Advanced; Exarafenib; binimetinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Neoplasm Metastasis; Thyroid Diseases | interventions — binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation Monotherapy (Part A1) (Experimental): Dose escalation of KIN-2787
  Interventions: Drug: KIN-2787
- Dose Escalation Combination therapy (Part A2) (Experimental): Dose escalation of KIN-2787 and binimetinib
  Interventions: Drug: KIN-2787 and binimetinib
- Dose Expansion Monotherapy (Part B1) (Experimental): Dose expansion evaluating the recommended phase 2 dose (RP2D) of KIN-2787
  Interventions: Drug: KIN-2787
- Dose Escalation Combination therapy (Part B2) (Experimental): Dose expansion evaluating the recommended phase 2 dose (RP2D) of KIN-2787 and binimetinib
  Interventions: Drug: KIN-2787 and binimetinib

INTERVENTIONS:
Drug: KIN-2787 — KIN-2787 will be administered orally twice daily in 28-day cycles
  Other Names: exarafenib
  Arms: Dose Escalation Monotherapy (Part A1); Dose Expansion Monotherapy (Part B1)
Drug: KIN-2787 and binimetinib — Continuous and Ramp-Up cohorts: KIN-2787 (exarafenib) and binimetinib will be administered orally twice daily in 28-day cycles Intermittent Cohort: KIN-2787 will be administered orally twice daily and binimetinib will be administered twice daily for 5 days on, 2 days off for 28-day cycles
  Other Names: exarafenib and binimetinib
  Arms: Dose Escalation Combination therapy (Part A2); Dose Escalation Combination therapy (Part B2)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of KIN-2787 in adults with BRAF/NRAS-mutated advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
This is a two-part, open-label, multi-center, dose escalation and dose expansion study in participants with BRAF mutation-positive and/or NRAS mutation-positive tumors designed to evaluate the safety, tolerability, and pharmacokinetics (PK) of KIN-2787, a RAF small molecule kinase inhibitor, to determine a recommended Phase 2 dose (RP2D) of KIN-2787, and to assess the objective response to KIN-2787 therapy alone and in combination with binimetinib, a mitogen-activated protein kinase (MEK) inhibitor.

The dose expansion phase (Part B) will assess the safety and efficacy of KIN-2787 at the recommended dose and schedule in patients with cancers that contain BRAF Class I, II or III mutations, including lung cancer, melanoma, and other selected solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to initiation of any study-specific procedures.
* Metastatic or advanced stage solid tumor
* Known BRAF Class I, Class II, or Class III alteration or melanoma with an NRAS mutation as confirmed by previous genomic analysis of tumor tissue or ctDNA.
* Measurable (Part A and B) or evaluable (Part A only) disease by RECIST v1.1.
* ECOG performance status 0-1
* Adequate organ function, as measured by laboratory values (criteria listed in protocol).
* Able to swallow, retain, and absorb oral medications.

Exclusion Criteria:

* Known participants who have received local therapy with either surgery and/or radiation therapy (participants with asymptomatic untreated brain metastasis may be eligible if met with certain criteria)
* In Part B Dose Expansion, previous treatment with any approved or in-development small molecule BRAF-, MEK-, or MAPK-directed inhibitor therapy.
* GI tract disease causing an inability to take oral medication, malabsorption syndrome, requirement for intravenous alimentation, or uncontrolled inflammatory GI disease.
* Active, uncontrolled bacterial, fungal, or viral infection.
* Participant with a positive test result for SARS-CoV2 infection, is known to have asymptomatic infection or is suspected of having SARS-CoV2, is excluded
* Women who are lactating or breastfeeding, or pregnant.
* Participants with any other active treated malignancy within 3 years prior to enrollment

Complete inclusion and exclusion criteria are listed in the clinical study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Part A1 Dose escalation monotherapy: | Initiation of study drug through 28 days after last dose (up to approximately 18 months)
  To determine the safety and tolerability of oral administration of KIN-2787 including dose-limiting toxicities (DLTs), and to identify the maximum tolerated dose (MTD) and/or the appropriate dose for further clinical investigation in Part B Dose Expansion.
Part A2 Dose Escalation: KIN-2787 + Binimetinib Combination | Initiation of study drug through 28 days after last dose (up to approximately 18 months)
  To determine the safety and tolerability of oral administration of KIN-2787 + binimetinib including DLTs, and to identify the MTD and/or the appropriate dose for further clinical investigation.
In Part B (Dose Expansion) - objective response rate (ORR) using RECIST v1.1. | Initiation of study drug until disease progression (up to approximately 36 months)
  To assess preliminary evidence of the anti-cancer activity of KIN-2787 and for (B2) KIN-2787 + binimetinib
In Part B (Dose Expansion) - disease control rate (DCR). | Initiation of study drug until disease progression (up to approximately 36 months)
In Part B (Dose Expansion) - duration of overall response (DOR). | Initiation of study drug until disease progression (up to approximately 36 months)
  Measure of clinical benefit, defined as the time from initial tumor response to documented tumor progression
In Part B (Dose Expansion) - duration of stable disease. | Initiation of study drug until disease progression (up to approximately 36 months)

SECONDARY OUTCOMES:
Part A1 Dose Escalation: Characterization of PK properties and effect of food on PK of KIN-2787 including, but not limited to tmax. | Initiation of study drug through Cycle 5, where each cycle is 28 days (up to approximately 4 months)
Part A1 Dose Escalation: Characterization of PK properties and effect of food on PK of KIN-2787 including, but not limited to AUC. | Initiation of study drug through Cycle 5, where each cycle is 28 days (up to approximately 4 months)
Part A1 Dose Escalation: Characterization of PK properties and effect of food on PK of KIN-2787 including, but not limited to Cmax. | Initiation of study drug through Cycle 5, where each cycle is 28 days (up to approximately 4 months)
Part A2 Dose Escalation: characterization of PK properties of KIN-2787 and binimetinib in combination including, but not limited to Cmax. | Initiation of study drug through Cycle 5, where each cycle is 28 days (up to approximately 4 months)
Part A2 Dose Escalation: characterization of PK properties of KIN-2787 and binimetinib in combination including, but not limited to AUC. | Initiation of study drug through Cycle 5, where each cycle is 28 days (up to approximately 4 months)
Part A2 Dose Escalation: characterization of PK properties of KIN-2787 and binimetinib in combination including, but not limited to tmax. | Initiation of study drug through Cycle 5, where each cycle is 28 days (up to approximately 4 months)
Part B Dose Expansion: characterization of PK properties of KIN-2787, and for (B2) KIN-2787 + binimetinib including, but not limited to AUC. | Initiation of study drug through Cycle 5, where each cycle is 28 days (up to approximately 4 months)
Part B Dose Expansion: characterization of PK properties of KIN-2787, and for (B2) KIN-2787 + binimetinib including, but not limited to Cmax. | Initiation of study drug through Cycle 5, where each cycle is 28 days (up to approximately 4 months)
Part B Dose Expansion: characterization of PK properties of KIN-2787, and for (B2) KIN-2787 + binimetinib including, but not limited to tmax. | Initiation of study drug through Cycle 5, where each cycle is 28 days (up to approximately 4 months)

CONTACTS AND LOCATIONS:
Overall Officials: CLaire FABRE, MD, Study Chair — Pierre Fabre Laboratories
Locations (50):
- United States (17):
  - The Angeles Clinic, Los Angeles, California
  - UCLA, Los Angeles, California
  - University of California San Diego, Moores Cancer Center, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Sarah Cannon Research Institute Denver, Denver, Colorado
  - Mayo Clinic - Florida, Jacksonville, Florida
  - Sarah Cannon Research Institute - Florida Cancer Specialists, Orlando, Florida
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Atlantic Health, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Sarah Cannon Research Institute-Tennessee Oncology, Nashville, Tennessee
  - MD Anderson, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Australia (5):
  - Calvary Mater Hospital Newcastle, Waratah, New South Wales
  - Melanoma Institute Australia, Wollstonecraft, New South Wales
  - Tasman Health Care, Southport, Queensland
  - Austin Health, Heidelberg, Victoria
  - Linear Clinical Research, Perth, Western Australia
- China (4):
  - Harbin Medical University Cancer Hospital, Haerbin, Heilongjiang
  - Linyi Cancer Hospital, Linyi, Shandong
  - Beijing University Cancer Hospital, Beijing
  - The Shanghai Pulmonary Hospital, Shanghai
- France (12):
  - Institut Bergonie, Bordeaux
  - Centre Francois Baclesse, Caen
  - CHU de Lille, Lille
  - Centre Leon Berard, Lyon
  - APHM-CHU La Timone, Marseille
  - CHU Nantes-Hotel Dieu, Nantes
  - CHU de Nice - Hôpital Archet 2, Nice
  - APHP - Hôpital St Louis, Paris
  - Hospices Civiles de Lyon - Hôpital Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Oncopole Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- Istituto Nazionale dei Tumori Fondazione G. Pascale, Napoli, Italy
- Spain (10):
  - Arance, Barcelona, Spain
  - NEXT Quirónsalud Madrid, Madrid, Spain
  - H. Regional de Málaga, Málaga, Spain
  - H. Virgen Macarena, Seville, Spain
  - Berrocal, Valencia, Spain
  - Hospital Quiron Dexeus, Barcelona
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria
  - START Madrid, Madrid
  - Hospital General Gregorio Marañón, Madrid
  - INCLIVA (Hospital Clinico de Valencia), Valencia
- National Taiwan University Hospital, Taipei, Taiwan